CLINICAL TRIAL: NCT02356458
Title: Combination of Ibrutinib and Bortezomib Followed by Ibrutinib Maintenance to Treat Patients With Relapsed and Refractory Mantle Cell Lymphoma; a Multicenter Phase I/II Trial.
Brief Title: Combination of Ibrutinib and Bortezomib to Treat Patients With Mantle Cell Lymphoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: SAKK Board decision of 14th November 2020 due to financial reasons.
Sponsor: Swiss Cancer Institute (Other)
Collaborators: European Mantle Cell Lymphoma Network (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 36/13; 2014-003893-17 (EudraCT Number); SNCTP000001235 (Other: Swiss National Clinical Trial Portal)
Record Dates: First submitted 2015-02-02; First posted 2015-02-05 (Estimated); Last update posted 2022-03-11 (Actual); Status verified 2022-02

CONDITIONS: Mantle Cell Lymphoma
Keywords: Mantle cell lymphoma; Relapsed; Refractory; Cancer; Lymphoma; Ibrutinib Imbruvica; Bortezomib Velcade
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Recurrence; Neoplasms; Lymphoma | interventions — ibrutinib; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ibrutinib & Bortezomib (Experimental): Combination therapy (trial treatment of ibrutinib in combination with bortezomib) followed by ibrutinib maintenance therapy
  Interventions: Drug: Ibrutinib; Drug: bortezomib

INTERVENTIONS:
Drug: Ibrutinib — Combination therapy:
  Trial treatment of ibrutinib in combination with bortezomib Cycles 1-6 (1 cycle = 21 days) Ibrutinib: p.o daily; Phase I: according to DL; Phase II: RP2D established in phase I
  Maintenance therapy:
  p.o daily: 560 mg
  Other Names: Imbruvica
Drug: bortezomib — Combination therapy:
  Trial treatment of ibrutinib in combination with bortezomib Cycles 1-6 (1 cycle = 21 days) Injection of Bortezomib (s.c.), dose of 1.3 mg/m2 on day 1, 4, 8, 11
  Other Names: Velcade®

SUMMARY:
Mantle cell lymphoma (MCL) remains an incurable disease with frequent relapses and no standard therapeutic options in case of relapse. Prolongation of remissions or induction of longer remissions is therefore crucial. Recently, a synergistic increase in the proteasomal inhibition of ibrutinib in both bortezomib-sensitive and refractory MCL cells was shown. These findings, along with the reported single agent activities of both drugs and the non-overlapping toxicities, are the rationale to combine ibrutinib and bortezomib in MCL in this trial

DETAILED DESCRIPTION:
Disease background, therapy background and aim

Mantle cell lymphoma (MCL) is a distinct subtype of B-cell lymphoma. It represents ~5% of all lymphomas and typically is present in advanced stages, a median age of 60-65 years and a dismal prognosis with a median survival of ~3 years. Currently, it remains incurable, as the patients will relapse after first line treatment and require subsequent therapy. The disease-free survival is progressively shorter with each subsequent relapse.

Currently, there is no standard therapy for relapsed MCL patients. MCL is predominantly a disease of the elderly who are not suitable for aggressive chemotherapy. Allogeneic transplants are preferred in young and fit patients, whereas (preferably single agent) chemotherapy is used to treat older patients, but usually with short duration of responses. Recently, the therapeutic armamentarium has been expanded with the availability of novel agents targeting crucial and deregulated pathways in MCL. These include the Bruton's Kinase (BTK) inhibitor ibrutinib with excellent single agent activities. New therapeutic options in the targeted patient population are clearly needed to prolong remissions especially for elderly patients where aggressive chemotherapy and allogeneic transplants are no suitable treatment options. Recently, a synergistic increase in the proteasomal inhibition of ibrutinib in both bortezomib-sensitive and refractory MCL cells was shown.

This trial is targeting patients with diagnosis of refractory or relapsed MCL disease after pretreatment with ≤2 lines of non-bortezomib-containing chemotherapy. The proposed treatment of ibrutinib in combination with bortezomib might lead to an improvement of the therapy in the targeted relapsed/refractory patient population. Given the absence of a dose-limiting toxicity also when applied long-term, ibrutinib is well suited in this patient population as a maintenance therapy. Therefore, the combination treatment of the trial is followed by a maintenance therapy part for patients that had no disease progression. New treatment options should control the disease as best and long as possible.

Treatment

Treatment consists of 6 cycles of 21 days each of ibrutinib in combination with bortezomib, followed by a maintenance therapy with ibrutinib monotherapy. In the maintenance therapy courses repeat every 28-days in the absence of disease progression or unacceptable toxicity.

Objectives Phase I The primary object of the trial is to establish the recommended phase II dose (RP2D) of ibrutinib in combination with bortezomib in patients with relapsed or refractory MCL.

The secondary objectives are

* to determine the safety and tolerability of ibrutinib in combination with bortezomib and
* to assess the preliminary antitumor activity of ibrutinib in combination with bortezomib Phase II The main object of the trial is to define the efficacy of the combination treatment of ibrutinib with bortezomib in patients with relapsed or refractory MCL.

The secondary objectives are

* to determine the safety and tolerability of the RP2D and
* to assess the efficacy of ibrutinib in combination with bortezomib in patients with relapsed MCL followed by an ibrutinib maintenance therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient must give written informed consent before registration indicating that the patient understands the purpose of the procedures required for the trial and is willing to participate in the trial.
* Histologically confirmed mantle cell lymphoma with either overexpression of cyclin D1 protein or evidence of t(11;14)(q13;q32) assessed by cytogenetics, by fluorescence, in situ hybridization (FISH) or by polymerase chain reaction (PCR).
* Refractory or relapsed disease in need of systemic therapy after pretreatment with non-bortezomib-containing chemotherapy (including high-dose therapy)
* At least one measurable lesion ≥11 mm in its greatest transverse diameter measured with CT scan (contrast enhanced) or MRI (in case of the disease cannot be adequately imaged using CT and if contrast is not appropriate for patients according to the treating physician)
* WHO performance status 0-2
* Age ≥ 18 years
* Adequate hematological values:

  * Absolute neutrophil count (ANC) > 1.0 x 109/L independent of growth factor support
  * Platelets ≥ 100 x 109/L or ≥ 50 x 109/L if bone marrow involvement independent of transfusion support in either situation,
  * Hb ≥ 80 g/L
* Adequate hepatic function:

  * Total bilirubin ≤1.5xupper limit of normal (ULN) unless bilirubin is due to Gilbert's syndrome ≤ 5.0 x ULN
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3xULN
* Adequate renal function: Body surface area (BSA) corrected creatinine clearance >40mL/min/1.73m2 (calculated according to the formula of Cockcroft-Gault)
* Women of childbearing potential and men who are sexually active must be practicing a highly effective method of birth control during and after the trial (see below) consistent with local regulations regarding the use of birth control methods for patients participating in clinical trials (see section 9.12). Men must agree to not donate sperm during and after the trial. These restrictions apply for

  * Ibrutinib: 3 month after the last dose of trial drug for males and 1 month for females.
  * Bortezomib: during trial treatment (for males and females): no restrictions of birth control after last dose of trial drug. Donation of sperm: 6 month after the last dose of trial drug.
* Women of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [β-hCG]) or urine pregnancy test at baseline. Women who are pregnant or breastfeeding are ineligible for this trial.

Exclusion Criteria:

* Prior therapy with ibrutinib or bortezomib
* Adverse event neuropathy of prior therapy grade ≥2 (according to CTCAE criteria) at registration
* Previous malignancy within 5 years with the exception of adequately treated in situ cervical cancer or localized non-melanoma skin cancer.
* Presence or history of CNS disease (either CNS lymphoma or lymphomatous meningeosis)
* Evidence of ongoing systemic infections of all kind
* Exclusion of the following prior treatments prior to trial registration

  * major surgery within 4 weeks
  * concurrent treatment with other experimental drugs or treatment in a clinical trial within 30 days.
  * treatment with chemotherapy and radiotherapy within ≥ 3 weeks
  * vaccinated with live, attenuated vaccines within 4 weeks
* History of stroke or intracranial hemorrhage within 6 months prior to trial registration.
* Requires anticoagulation with warfarin or equivalent vitamin K antagonists (e.g. phenprocoumon)
* Requires treatment with strong or moderate CYP3A inhibitors (see http://medicine.iupui.edu/)
* Clinically significant cardiovascular disease such as congestive heart failure NYHA III or IV (as defined by the New York Heart Association Functional Classification), uncontrolled or symptomatic arrhythmias, significant QT-prolongation, unstable angina pectoris myocardial infarction within 6 months of prior to registration,
* Known history of human immunodeficiency virus (HIV) or active Hepatitis C virus or active Hepatitis B virus infection or any uncontrolled active systemic infection requiring treatment.
* Prior allogeneic bone marrow or solid organ transplantation
* Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion,

  * could impair the ability of the patient to participate in the trial
  * could compromise the patient's safety,
  * could interfere with the absorption or metabolism of ibrutinib capsules, or
  * could put the trial outcomes at undue risk
  * could prevent compliance with trial treatment.
* Psychiatric disorder precluding understanding of trial information, giving informed consent, or interfering with compliance for oral drug intake.
* Known hypersensitivity to trial drug(s) or hypersensitivity to any other component of the trial drugs.
* Any concomitant drugs contraindicated for use with the trial drugs according to the approved product information.
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the trial protocol and follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2015-08-31 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Phase I: Dose limiting toxicity (DLT) observed during the first cycle of trial treatment | At day 8, 14, 21 during cycle 1 (1 cycle = 21 days)
  DLTs are defined based on adverse events observed in cycle 1 that are possibly, probably or definitively related to ibrutinib and/or bortezomib.
Phase II: Overall response (OR) (combination therapy) | 4 1/2 months after registration.
  OR is defined as the proportion of patients whose best overall response, is either complete response (CR), complete response unconfirmed (CRu) or partial response (PR) according to the International Working group criteria for NHL. The primary endpoint of phase II is OR observed during the combination therapy.

OTHER OUTCOMES:
Phase I and II: Adverse events (AE) until 30 days after end of trial therapy | Until 30 days after up to 2 years of trial therapy
  All AEs will be assessed according to NCI CTCAE v4.0
Phase I: OR (combination therapy) | 4 1/2 months after inclusion of each patient
  OR observed during the combination therapy.
Phase I: OR based on best response observed during treatment (combination and maintenance therapy) | Estimated at 1 1/2 years after patient registration.
  OR observed during the combination therapy and OR observed during trial treatment.
Phase II: OR based on best response observed during treatment (combination and maintenance therapy | Estimated at 1 1/2 years after patient registration.
  OR observed during the combination therapy and OR observed during trial treatment.
Phase II: Progression-free survival (PFS) | Time from patient registration to progression free survival (estimated 2 years)
  Time from registration until progression of disease or death as a result of any cause.
Phase II: Time to treatment failure (TTF) | Time from patient registration to treatment failure (estimated 2 years)
  Time from registration until treatment failure (due to unacceptable toxicity, progression, patient refusal, death, start of subsequent anti-MCL therapy or any other event that determines the termination of the trial treatment will be considered as treatment failure).
Phase II: Duration of objective response | Time from patient registration to progression/relapse (estimated 2 years).
  Time from first observation of CR or PR until documentation of progression, or relapse thereafter.
  Only patients with CR or a PR will be included in this analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Urban Novak, PD Dr. med., Study Chair — University Hospital Bern - Inselspital
Locations (19):
- Germany (3):
  - Universitätsmedizin Mainz, Mainz
  - Klinikum der Universität München, München
  - Universitätsmedizin Rostock, Rostock
- Italy (3):
  - Azienda Ospedaliera SS Antonio e Biagio e Cesare Arrigo, Alessandria
  - European Institute of Oncology, Milan
  - Università di Torino, Torino
- Switzerland (13):
  - Kantonsspital Aarau, Aarau
  - Kantonsspital Baden, Baden
  - Inselspital, Bern, Bern
  - Kantonsspital Graubünden, Chur
  - Hopitaux Universitaires de Geneve, Geneva
  - Centre Pluridisciplinaire d'Oncologie CHUV, Lausanne
  - Kantonsspital Baselland, Liestal
  - Istituto Oncologico della Svizzera Italiana, Lugano
  - Kantonsspital Luzern, Luzerne
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Onkozentrum - Klinik Im Park, Zurich
  - UniversitätsSpital Zürich, Zurich
  - Klinik Hirslanden, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Novak U, Fehr M, Schar S, Dreyling M, Schmidt C, Derenzini E, Zander T, Hess G, Mey U, Ferrero S, Mach N, Boccomini C, Bottcher S, Voegeli M, Cairoli A, Ivanova VS, Menter T, Dirnhofer S, Scheibe B, Gadient S, Eckhardt K, Zucca E, Driessen C, Renner C. Combined therapy with ibrutinib and bortezomib followed by ibrutinib maintenance in relapsed or refractory mantle cell lymphoma and high-risk features: a phase 1/2 trial of the European MCL network (SAKK 36/13). EClinicalMedicine. 2023 Sep 22;64:102221. doi: 10.1016/j.eclinm.2023.102221. eCollection 2023 Oct. PMID 37781158